CLINICAL TRIAL: NCT02441023
Title: Nutritional Therapy and Education With a Multimedia Application in the Metabolic Control of Patients With Type 2 Diabetes. Randomized Clinical Trial
Brief Title: Nutritional Therapy and Education With Multimedia Application in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Lubia Velázquez López, M.Cs, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-C01-181015
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes mellitus; nutritional therapy; health education; self-management; multimedia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Education | interventions — Nutrition Therapy; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional therapy and education (Experimental): 1. Nutritional therapy guidance according to sex, age, weight and comorbidity present. The recommendations of calories and macronutrients intake were indicated according to the Official Mexican Standards for Diabetes treatment and the American Diabetes Association standards for medical care in diabetes.
  2. Education with multimedia application: Patients were exposed to the multimedia application previous to the nutritional counseling. Multimedia application comprises the following modules: 1) Introduction, 2) Nutrition, 3) Physical Exercise, 4) Diabetes myths 5) Metabolic control indicators 6) Knowing diabetes, 7) Diabetes complications including testimonials.
  Interventions: Behavioral: Nutritional therapy and education; Behavioral: Nutritional therapy
- Nutritional Therapy (No Intervention): Nutritional therapy guidance according to sex, age, weight and comorbidity present. The recommendations of calories and macronutrients intake were indicated according to the Official Mexican Standards for Diabetes treatment and the American Diabetes Association standards for medical care in diabetes.

INTERVENTIONS:
Behavioral: Nutritional therapy and education — 1. Nutritional therapy guidance according to sex, age, weight and comorbidity present. The recommendations of calories and macronutrients intake were indicated according to the Official Mexican Standards for Diabetes treatment and the American Diabetes Association standards for medical care in diabetes.
  2. Education with multimedia application: Patients were exposed to the multimedia application previous to the nutritional counseling. Multimedia application comprises the following modules: 1) Introduction, 2) Nutrition, 3) Physical Exercise, 4) Diabetes myths 5) Metabolic control indicators 6) Knowing diabetes, 7) Diabetes complications including testimonials.
  Arms: Nutritional therapy and education
Behavioral: Nutritional therapy — Nutritional therapy guidance according to sex, age, weight and comorbidity present. The recommendations of calories and macronutrients intake were indicated according to the Official Mexican Standards for Diabetes treatment and the American Diabetes Association Standards for medical care in diabetes.
  Arms: Nutritional therapy and education

SUMMARY:
The purpose of this study is to evaluate the effectiveness of nutrition therapy in combination with education in diabetes using a multimedia application for improving indicators of metabolic control in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Randomized clinical trial. Subjects with type 2 diabetes from three Family Medicine Units (primary care), with HbA1c >6.5% and <13.0%, without advanced macro or microvascular complications of diabetes.

Two arms: the experimental group with nutrition therapy plus education in diabetes through a multimedia application. The application had seven modules: Introduction, nutrition, physical exercise in diabetes, myths and truths on diabetes, metabolic control parameters, knowing diabetes, complications of diabetes. The control group received only usual nutrition therapy.

A monthly follow up during the first 7 months and then bimonthly, until 21 months of total follow up, with reinforcement in each visit of nutrition and other non-pharmacological therapy, with control on weight and blood pressure. Laboratory studies included HbA1c, lipids profile, creatinine and albuminuria, performed at 7, 14 and 21 months. Results were provided to both the patient and his family physician, so modification in drug treatment if needed, were performed.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of type 2 diabetes, following ADA & WHO criteria
* Without severe marco or microvascular complications of diabetes
* HbA1c > 6.5% and <13.0%

Exclusion criteria:

* Inability to or unwillnigness to access the multimedia or to follow dietary recommendations

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Metabolic control | 21 months
  metabolic control which is evaluated by measuring the change in glycosylated hemoglobin

SECONDARY OUTCOMES:
Lipids profile | 21 months
  Lipid profile includes the evaluation of total cholesterol, triglycerides, HDL-c and LDL-c
Body mass index (BMI) | 21 months
  It is evaluated by measuring the weight in relation to height

CONTACTS AND LOCATIONS:
Overall Officials: Lubia Velazquez, M. Sc.,, Principal Investigator — Unidad de Investigación en Epidemiología Clínica, Hospital Regional Carlos Mac Gregor Sanchez Navarro, IMSS
Locations (1):
- Unidad de Investigación en Epidemiología Clínica, Hospital Regional 1 Carlos Mac Gregor Sanchez Navarro, IMSS, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Provide nutritional and educational measures in long-term in diabetes care.